CLINICAL TRIAL: NCT06216314
Title: Effects of Race Pace Based Approach on the Performance of Recreational Runners: a Randomized Controlled Trial
Brief Title: Effects of Race Pace Based Approach in Recreational Runners
Acronym: 22HUM23661
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Collaborators: GO fit Lab- Ingesport (Network)
Responsible Party: Principal Investigator, Arturo Casado, Principal Investigator, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1201202302023; 22HUM-23661 (Other Grant/Funding Number: Comunidad Autonoma de Madrid (CAM))
Record Dates: First submitted 2023-12-21; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Healthy
Keywords: heart rate variability; endurance training; HRV-guided; periodization; training intensity distribution
MeSH Terms: interventions — Heart Rate

STUDY DESIGN:
Intervention Model Description: A 4-week pre-intervention plus 6-week intervention program was set up. Participants were randomly assigned to one of the three groups before the intervention phase using a web-based computer program (www.randomizer.org).
  A randomized controlled trial with three-armed parallel group was set.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Heart rate (HR) (Active Comparator): Three physiological zones were established according to the results of the treadmill test. The HR group completed training sessions based on HR values and velocities associated with ventilatory thresholds (i.e., Z1, zone 1: intensity zone below the first ventilatory threshold; Z2: zone 2, intensity zone between the first and second ventilatory threshold; Z3: zone 3, intensity zone above the second ventilatory threshold. Runners trained 4 times a week.
  Interventions: Other: Heart rate (HR)
- Race pace based approach (RP) (Experimental): For the race pace based approach (RP), intensity zones were established by calculating the percentage of the average speed achieved in the 7-km time trial (TT) and 3 zones were established. Kenneally's model was used to determine the race intensity zones by analyzing 7-km TT performance. Z1 corresponds to less than 80% of race pace, Z2 is between 80-95%, and Z3 corresponds to over 95% of race pace. Runners trained 4 times a week.
  Interventions: Other: Race pace based approach (RP)
- Heart rate + heart rate variability (HRV) (Experimental): The HR+HRV group completed training sessions based on HR values and velocities associated with ventilatory thresholds (i.e., Z1, zone 1: intensity zone below the first ventilatory threshold; Z2: zone 2, intensity zone between the first and second ventilatory threshold; Z3: zone 3, intensity zone above the second ventilatory threshold. The training sessions were based on physiological thresholds and daily HRV cues. Runners trained 4 times a week.
  Interventions: Other: Heart rate + heart rate variability (HRV)

INTERVENTIONS:
Other: Heart rate (HR) — Runners ran according to speeds and HR associated with ventilatory thresholds. Z1, zone 1: intensity zone below the first ventilatory threshold; Z2: zone 2, intensity zone between the first and second ventilatory threshold; Z3: zone 3, intensity zone above the second ventilatory threshold.
  Other Names: HR
  Arms: Heart rate (HR)
Other: Race pace based approach (RP) — Runners ran respecting three intensity zones.
  The average speed achieved in the 7-km was calculated. From this, three intensity zones were calculated, adhering to the % of the race pace of the 7-km test.
  Z1 corresponds to less than 80% of race pace, Z2 is between 80-95%, and Z3 corresponds to over 95% of race pace
  Other Names: RP
  Arms: Race pace based approach (RP)
Other: Heart rate + heart rate variability (HRV) — Runners completed training sessions based on HR values and velocities associated with ventilatory thresholds (i.e., Z1, zone 1: intensity zone below the first ventilatory threshold; Z2: zone 2, intensity zone between the first and second ventilatory threshold; Z3: zone 3, intensity zone above the second ventilatory threshold. The training sessions were based on physiological thresholds and daily HRV cues. High-intensity training was performed only under optimal HRV conditions, thus only when each participant had HRV values in their reference range. If HRV was not optimal, low-intensity training was prescribed. If HRV was not optimal for two days consecutively, rest was prescribed.
  Other Names: HR+HRV
  Arms: Heart rate + heart rate variability (HRV)

SUMMARY:
The aim of the study was to compare the performance effects of the intensity demarcation model based on the race pace based approach with the triphasic physiological model and heart rate variability guidelines (HR+HRV)

DETAILED DESCRIPTION:
After being informed and signing informed consent about the present study, participants were randomly assigned to one of three groups before the intervention phase using a Web-based computer program (www.randomizer.org). Groups were matched on a 1:1:1 basis by gender, age, and performance in an official 10-km race in the previous month. Once selected, participants in the heart rate variability (HRV) group began daily measurements to obtain their personalized parameters.

The groups changed according to the intensity zone demarcation pattern: heart rate (HR), race pace (RP) and HR+HRV. The HR group was considered the active control group, as considered the current best practice according to the current literature in endurance running. A 4-week pre-intervention plus 6-week intervention program was set up.

Participants were assessed in four different sessions, two for laboratory evaluations and two for time trial performance. The first session consisted of a running economy test, and, after at least half an hour of rest, a maximal incremental treadmill run. They familiarised themselves with the training sessions according to their group (i.e., running based on HR, RP or HR+HRV guidelines, respectively).

The HRV4training mobile application (https://www.hrv4training.com) was used to assess HRV for one minute in the morning. The difference in RR intervals between heartbeats is used to calculate HRV. The program then uses this information to calculate the rMSSD and moving average (LnrMSSD7-d), converting the results to a number between 5 and 10. Then, the participant must answer a series of questions including his or her current physical state, sleep quality, muscle soreness, etc. After interpolating these variables, the application shows the subjective value derived from the body's reaction to stresses. As a result, daily indications are given in numerical form, with a range of normality (for HR and HRV) that varies each day depending on how the person reacts to stress. Participants were instructed to take the measurement as soon as they woke up, with an empty bladder, lying down, trying to limit movement, and breathing naturally

Training variables (total time, distance, total time spent in each zone) and Training Impulse (TRIMP) were the same for all groups

ELIGIBILITY:
Inclusion Criteria:

* Being adults
* VO2max between 45 and 60 mL·min-1·kg^-1 for men
* VO2max between 40 and 55 mL·min^-1 for women
* More than 4 days per week of training frequency
* Running experience ≥ 2 years
* Record HR data of all training sessions during the study

Exclusion Criteria:

* Previous injuries for at least three months
* Smokers
* Any cardiovascular condition that compromises health status and participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Change from Baseline of Running Economy | Baseline and after 6 weeks
  Tests were performed on the treadmill and respiratory gas analysis was carried out.
  The laboratory tests included:
  - Running economy (RE) test (ml·kg·km)
  RE was measured by running two blocks at constant speeds (7 and 9 km·h^-1 or 8 and 10 km·h^-1, respectively), depending on the subject's level, intensities below the first ventilatory threshold. Each block lasted three minutes.
  RE is one of the physiological determinants of endurance performance: an improvement in RE over time indicates an improvement in performance
Change from Baseline of VO2max | Baseline and after 6 weeks
  Tests were performed on the treadmill and respiratory gas analysis was carried out.
  The laboratory tests included:
  - Maximum oxygen consumption test (VO2max)
  After 30 minutes of rest, a maximal incremental test was performed to calculate relative VO2max (ml·kg^-1·min^-1) and absolute VO2max (L·min^-1).
  The test started at the last speed of the RE test (9 or 10 km·h^-1), depending on the subject's level. The speed increased continuously by 0.5 km·h-1 every minute until exhaustion. The mean value of the last 30 s of the VO2, a respiratory exchange ratio (RER) >1.05, a HR > 95% of the maximum HR, and an RPE > 18 were the variables considered to calculate the VO2max
  VO2max is one of the determinants of endurance performance. The relative VO2max is influenced by weight (at equal VO2max, the runner who weighs less is more advantaged). An improvement in absolute and relative values of VO2max over time indicate an improvement in performance
Change from Baseline of Maximum aerobic velocity (VAM) | Baseline and after 6 weeks
  Tests were performed on the treadmill and respiratory gas analysis was carried out.
  The laboratory tests included:
  - Maximum aerobic velocity (VAM) in km·h^-1
  VAM was calculated as the minimum speed that elicits maximum oxygen consumption.
  VAM is one of the physiological determinants of endurance performance. An increase in VAM velocity over time is an indication of improved performance
Change from Baseline of 7-km Time Trial Performance | Baseline and after 6 weeks
  Before and after 6 weeks, the final time achieved in a 7-km time trial performance was calculated for all participants.
  The athletes were instructed to achieve their best performance on the 7-km. The test was performed in a 400m regulation athletic track. Verbal encouragement was given to all runners in both tests every 400-m lap.
  Participants used the same shoe model in the two tests and were asked not to use stimulants (coffee, tea, etc.). They performed the tests at the same time of day ± (2 hours).
  A decrease in the final time in the second test, indicates an improvement in performance
Change from Baseline of the First Physiological Thresholds (VT1) | Baseline and after 6 weeks
  Ventilatory thresholds (VT1 and VT2), measured by gas analysis, are some of the determinants of endurance performance, along with running economy and VO2max.
  Were measured changes in:
  - Velocity associated with the first ventilatory threshold (VT1) in km·h^-1
  Velocity zones corresponding to VT1 indicates a low intensity zone. An increase over time in VT1 indicates an improvement of the aerobic system
Change from Baseline of the second Physiological Thresholds (VT2) | Baseline and after 6 weeks
  Ventilatory thresholds (VT), measured by gas analysis, are some of the determinants of endurance performance, along with running economy and VO2max.
  Were measured changes in:
  - Velocity associated with the second ventilatory threshold (VT2) in km·h^-1.
  Intensity zones corresponding to VT2 indicates a high intensity zone. An increase over time in VT2 indicates an improvement in the anaerobic system
Change from baseline in HR associated with the first ventilatory threshold | Baseline and after 6 weeks
  Ventilatory thresholds (VT), measured by gas analysis, are some of the determinants of endurance performance, along with running economy and VO2max.
  were measured changes in:
  - HR associated with the first ventilatory threshold HR-VT1 in beats per minute (bpm).
  A lower HR associated with VT1, indicates an improvement of the aerobic system over time
Change from baseline in HR associated with the second ventilatory threshold | Baseline and after 6 weeks
  Ventilatory thresholds (VT), measured by gas analysis, are some of the determinants of endurance performance, along with running economy and VO2max.
  were measured changes in:
  - HR associated with the second ventilatory threshold (HR-VT12) in beats per minute (bpm).
  Higher HR associated with VT2, indicates an improvement of the anaerobic system over time

SECONDARY OUTCOMES:
Change of Rate of Perceived Exertion (RPE) scale after 6 weeks protocol | Baseline and after 6 weeks
  Participants indicated Rating of perceived exertion (RPE) using Borg's 6-20 validated scale, an exertion perception scale used during laboratory testing. RPE values were measured for both the running economy and during the incremental maximal test (VO2max).
  The RPE values are:
  6. = no exertion at all 7. = extremely light 9. = very light 11. = light 13. = somewhat hard 15. = hard (heavy) 17. = very hard 19. = extremely hard A decrease in RPE over time for the same intensity (e.g., same speed achieved in tests) indicates better performance adaptation
Changes in Body Weight | Baseline and after 6 weeks
  Participants were weighed before and after the study to calculate body composition analysis. Participants arrived well hydrated, and were instructed to eat at least two hours beforehand. Weighing was performed at the same time slot (± 2 hours).
  it was measured:
  - Body weight (kg)
Changes in Height (cm) | Baseline and after 6 weeks
  Participants were weighed before and after the study to calculate body composition analysis.
  Participants arrived well hydrated, and were instructed to eat at least two hours beforehand. Weighing was performed at the same time slot (± 2 hours).
  it was measured:
  - Height (cm)
Changes in BMI (kg/m^2) | Baseline and after 6 weeks
  Participants were weighed before and after the study to calculate body composition analysis:
  Participants arrived well hydrated, and were instructed to eat at least two hours beforehand. Weighing was performed at the same time slot (± 2 hours).
  it was measured:
  - BMI (kg/m^2)
Changes in Fat mass | Baseline and after 6 weeks
  Participants were weighed before and after the study to calculate body composition analysis:
  Participants arrived well hydrated, and were instructed to eat at least two hours beforehand. Weighing was performed at the same time slot (± 2 hours).
  it was measured:
  - Fat mass (%)
Changes in Free Fat Mass | Baseline and after 6 weeks
  Participants were weighed before and after the study to calculate body composition analysis:
  Participants arrived well hydrated, and were instructed to eat at least two hours beforehand. Weighing was performed at the same time slot (± 2 hours).
  it was measured:
  - Free fat mass (%)

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Casado, PhD, Principal Investigator — Centro de Investigación en Ciencias del Deporte; Alfonso Jiménez Gutiérrez, PhD, Study Director — Director del Centro de Investigación en Ciencias del Deporte
Locations (1):
- Universidad Rey Juan Carlos, Fuenlabrada, Madrid, Spain

REFERENCES:
- [Background] Carrasco-Poyatos M, Gonzalez-Quilez A, Martinez-Gonzalez-Moro I, Granero-Gallegos A. HRV-Guided Training for Professional Endurance Athletes: A Protocol for a Cluster-Randomized Controlled Trial. Int J Environ Res Public Health. 2020 Jul 29;17(15):5465. doi: 10.3390/ijerph17155465. PMID 32751204
- [Derived] Ranieri LE, Casado A, Martin D, Trujillo-Colmena D, Gil-Arias A, Kenneally M, Jimenez A. Performance and Physiological Effects of Race Pace-Based Versus Heart Rate Variability-Guided Training Prescription in Runners. Med Sci Sports Exerc. 2025 Jul 1;57(7):1510-1522. doi: 10.1249/MSS.0000000000003671. Epub 2025 Feb 12. PMID 39935030